CLINICAL TRIAL: NCT01533168
Title: Next-Generation Sequencing of Immunoglobulin Heavy Chain Variable Region to Identify Previously Undetectable Minimal Residual Disease in Children With Acute Lymphoblastic Leukemia With Prognostic Significance
Brief Title: Genetic Test To Identify Previously Undetectable Minimal Residual Disease in Cell Samples From Younger Patients With Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL12B1; COG-AALL12B1; CDR0000724799; AALL12B1 (Other: COG); NCI-2012-00246 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-09; First posted 2012-02-15 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cytogenetic Analysis; Base Sequence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — cell samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: cytogenetic analysis
Genetic: nucleic acid sequencing
Other: diagnostic laboratory biomarker analysis
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Testing for minimal residual disease in cell samples from patients with acute lymphoblastic leukemia may help doctors plan better treatment.

PURPOSE: This research trial studies a genetic test in identifying previously undetectable minimal residual disease in cell samples from younger patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify and characterize changes in clonal populations of B cells in children with acute lymphoblastic leukemia (ALL) at diagnosis and Day 29 of induction.
* To define the ability of this technology to reclassify patients as minimal residual disease (MRD) positive at Day 29 of induction.
* To determine whether more sensitive detection of MRD at Day 29 would have clinical prognostic value in children with ALL.

OUTLINE: DNA extracted from diagnostic cells are analyzed for immunoglobulin heavy chain variable region by next-generation sequencing.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Samples from patients enrolled on COG-AALL0232 with standard-risk (SR) or high-risk (HR) acute lymphoblastic leukemia (ALL) with varying levels of MRD and relapse
* Diagnostic cells and Day 29 cells from patients that have not relapsed and are 5 years from diagnosis on protocol COG-AALL0232
* Diagnostic cells and Day 29 cells from patients that are matched for age, sex, initial white blood cell (WBC) count, and cytogenetics that have relapsed

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients With Acute Lymphoblastic Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Identification and characterization of changes in clonal populations of B cells in children with ALL
Reclassification of patients as MRD positive at day 29
Higher sensitivity detection that allow the stratification of the MRD population into 2 groups with lower and higher likelihood of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Norman J. Lacayo, MD, Principal Investigator — Stanford University